CLINICAL TRIAL: NCT05424393
Title: Long-term Real-world Prospectiv Observational Study on Maintenance Treatment With YISAIPU, an Etanercept Biosimilar, for Patients Wih Rheumatoid Arthritis of Fujian Province of China
Brief Title: Real-World Study on Long-term Treatment With YISAIPU for Fujian RA Patients
Acronym: LORMYF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: FJ_RA_RWS_2021
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-03

CONDITIONS: Rheumatoid Arthritis
Keywords: clincal remission; low disease activity
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — no need
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RA Patients receiving routine treatment: During the induction phase, the dose of YISAIPU is 50mg/wk. Patients who achieved clinical remission or low activity after 24 weeks of induction treatment can enter the maintenance phase. Those who fail to succeed in induction treatment will not be followed up. During the maintenance phase, the dose of YISAIPU could be either 50mg/wk or 25mg/wk. Patients will be followed up regularly for 2.5 years.
  Interventions: Drug: YISAIPU® ( An etanercept biosimilar); Drug: csDMARDs

INTERVENTIONS:
Drug: YISAIPU® ( An etanercept biosimilar) — YISAIPU®, an etanercept biosimilar produced by 3SBio Inc., is a TNF-α inhibitor targeting soluble TNF-α to inhibit its interaction with cell-surface receptors. It has been widely used in clinical practice for 17 years in China. According to the prescription information, YISAIPU should be given as 25mg, biw, pc.
  Other Names: a recombinant tumor necrosis factor receptor-Fc fusion protein; rhTNFR:Fc
Drug: csDMARDs — csDMARDs include methotrexate, sulfasalazine, hydroxychloroquine and leflunomide The use of csDMARDs complies with clinical routine practice and treatment strategy of treat-to-target.

SUMMARY:
Through real-world observation, understanding clinical efficacy and safety of treatment with YISAIPU (etanercept biosimilar) for RA patients of Fujian Province for three years

DETAILED DESCRIPTION:
This is a multi-center, prospective, real-world observational study. Patients who have completed 6 months of induction therapy (YISAIPU 50mg / week ± csDMARDs) and achieved clinical remission or low disease activity will be observed for 2.5 years. During the maintenance period, through full communication between doctors and patients, YISAIPU 50 mg/wk or YISAIPU 25 mg/wk will be chosen as maintenance treatment. The clinical efficacy evaluation parameters include DAS28, HAQ-DI, modified Sharp score, continuous medication rate, and the recurrence rate of rheumatoid arthritis. Drug safety evaluation will include the incidence of adverse drug reactions and adverse drug events, the incidence of serious adverse events, and the incidence of adverse events leading to the reduction or withdrawal of YISAIPU due to adverse events. Exploratory observations wil include: (1) the incidence, clinical characteristics and disease changes of Interstitial Lung Disease, (2) the baseline abnormal rate and 3-year change of carotid intima-media thickness.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Meet the ACR revised RA classification criteria(2010);
* Disease duration is more than or equal to 6 weeks;
* DAS28-CRP>2.6;
* Patient is eligible for TNF inhibitors treatment according to the judgment of the attending doctor in clinical practice;
* A written informed consent form must be provided with a signed and signed date prior to the commencement of any study specific procedure.

Exclusion Criteria:

Exclusion criteria:

* Patient has contraindication(s) to the use of fusion-protein type of TNF inhibitor;
* Patient is participating in other ongoing drug clinical trials;
* Patient whose LTBI screening result is positive, or had not received standard anti-TB treatment for TB history, is unwilling to take prophylactic treatment for TB;
* Patient with HBV infection and positive for HBV replication (not up to active replication) is not willing to receive anti-HBV treatment;
* Anti-HCV antibody is positive and HCV-RNA is positive, and patient is unwilling to start anti-HCV treatment;
* Other reasons the researchers think the patient is not eligible for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients in routine clinical practice environments
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical remission defined by DAS28 | 48 weeks
  Clinical efficacy: Clinical remission rate achieved at 48 weeks

SECONDARY OUTCOMES:
clinical remission rate of RA at weeks 24, 96 and 144 | weeks 24, 96 and 144
  clinical remission rate of RA at weeks 24, 96 and 144
low disease activity rate of RA at weeks 24, 48, 96 and 144 | weeks 24, 48, 96 and 144
  low disease activity rate of RA at weeks 24, 48, 96 and 144
joint function remission (HAQ ≤0.5) rate at weeks 24, 48, 96 and 144 | weeks 24, 48, 96 and 144
  joint function remission (HAQ ≤0.5) rate at weeks 24, 48, 96 and 144
improvement of radiographic progression of both hands evaluated by modified SHARP score at weeks 96 and 144 | weeks 24, 48, 96 and 144
  improvement of radiographic progression of both hands evaluated by modified SHARP score at weeks 96 and 144
scores of synovitis and bone erosion evaluated by ultrasound at week 24, 48, 96 and 144 | weeks 24, 48, 96 and 144
  scores of synovitis and bone erosion evaluated by ultrasound at week 24, 48, 96 ，144
rates of severe adverse reactions rate and severe adverse events at week 24, 48, 96 and 144 | weeks 24, 48, 96 and 144
  rates of severe adverse reactions rate and severe adverse events at week 24, 48, 96 and 144
changes of carotid intima-media thickness at weeks 48 and 144 | weeks 48 and 144
  changes of carotid intima-media thickness at weeks 48 and 144

CONTACTS AND LOCATIONS:
Overall Officials: Guixiu Shi, MD PHD, Study Director — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
share the study protocol
Supporting Information: Study Protocol
Time Frame: until completed
Access Criteria: Scholars in rheumatism